CLINICAL TRIAL: NCT01664156
Title: Effect of Korean Red Ginseng on Women With Cold Hypersensitivity of Hands and Feet : a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Korean Red Ginseng on Women With Cold Hypersensitivity of Hands and Feet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, JIN-MOO LEE, Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2012-004
Record Dates: First submitted 2012-08-08; First posted 2012-08-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Cold Hypersensitivity
Keywords: Cold hypersensitivity; Korean red ginseng; Infrared thermography; Cold stress test; Distal-dorsal difference
MeSH Terms: conditions — Cold Hypersensitivity | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Korean red ginseng (Experimental): The patients will receive Korean red ginseng(Korean Red Ginseng Powder Capsule®; Korea Ginseng Corporation, Daejeon, Korea). Patients will be requested to take 6 capsules 2 times a day (1h after breakfast and dinner).
  Interventions: Drug: Korean red ginseng
- placebo (Placebo Comparator): Placebo Korean red ginseng capsule contain cornstarch powder with the same color and taste as Korean red ginseng. Patients will be requested to take 6 capsules 2 times a day (1h after breakfast and dinner).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Korean red ginseng — Korean red ginseng is a steamed form of Panax ginseng with preserved major constituents. It has been shown to possess more biological activity than panax ginseng.
  Arms: Korean red ginseng
Drug: Placebo
  Arms: placebo

SUMMARY:
1. Objectives

   1. to verify effect of Korean red ginseng on cold hypersensitivity of hands and feet in women
   2. to establish scientific evidence for the use of Korean red ginseng by investigating changes of infrared thermography
2. Hypothesis The hypothesis is that Korean red ginseng will reduce cold hypersensitivity of hands and feet more effectively than placebo after 8 weeks administration of interventions- Korean red ginseng or the placebo.

DETAILED DESCRIPTION:
Design

* This trial is a randomized, double blind, placebo controlled trial with 80 patients.
* The trial will be implemented at Kyung Hee University Hospital at Gangdong in Seoul, Korea.
* Participants will take Korean red ginseng or placebo for 8 weeks and will be followed up during 4 weeks.
* During the administration period, 6 capsules 2 times a day (1h after breakfast and dinner) of Korean red ginseng or its placebo will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 16 to 60 years
2. Women complaining cold hypersensitivity on hands and feet
3. Thermal deviation between the palm and the upper arm is higher than 0.3℃

Exclusion Criteria:

1. Skin ailment, radiculopathy, thrombophlebitis, and injuries affecting infrared thermography
2. Alcohol abuse and alcoholic
3. History of cancer within 5 years
4. Severe depression
5. Hypertension and diabetes
6. Pregnancy or breastfeeding
7. Abnormal finding from blood test at screening visit
8. Allergic to Korean red ginseng
9. Took herbal medicine or health functional food within a week Participated another clinical trials within 3 months

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The change of the infrared thermography of cold hypersensitivity on hands | baseline and 8 weeks

SECONDARY OUTCOMES:
The change of the infrared thermography of cold hypersensitivity on feet | baseline and 8 weeks
The change of the Visual Analogue Scale of cold hypersensitivity on hands and feet | baseline and 8 weeks
The change of cold stress test | baseline and 8 weeks
The change of Distal-Dorsal Difference | baseline and 8 weeks
The change of Heart Rate Variability | baseline and 8 weeks
The change of 36-Item Short Form Health Survey | baseline, 8 weeks, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JIN-MOO LEE, Ph. D, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu, South Korea

REFERENCES:
- [Background] Hur YM, Chae JH, Chung KW, Kim JJ, Jeong HU, Kim JW, Seo SY, Kim KS. Feeling of cold hands and feet is a highly heritable phenotype. Twin Res Hum Genet. 2012 Apr;15(2):166-9. doi: 10.1375/twin.15.2.166. PMID 22856358
- [Derived] Park KS, Kim JW, Jo JY, Hwang DS, Lee CH, Jang JB, Lee KS, Yeo I, Lee JM. Effect of Korean red ginseng on cold hypersensitivity in the hands and feet: study protocol for a randomized controlled trial. Trials. 2013 Dec 19;14:438. doi: 10.1186/1745-6215-14-438. PMID 24354675